CLINICAL TRIAL: NCT01828944
Title: Olive Oil Polyphenols, Vitamin D and Docosahexaenoic Acid (DHA) Synergistic Effects on Locomotor Function
Brief Title: Olive Oil Polyphenols, Vitamin D, Docosahexaenoic Acid (DHA) and Locomotor Function (PolivD3)
Acronym: PolivD3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lesieur (Industry)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AU961; 2012-A00344-39 [N°IDRCB] (Other: French Health Agency)
Record Dates: First submitted 2013-04-02; First posted 2013-04-11 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-01

CONDITIONS: Osteopenia; Sarcopenia
Keywords: Vitamin D; bone loss
MeSH Terms: conditions — Bone Diseases, Metabolic; Sarcopenia | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Extra virgin olive oil (Active Comparator): Extra virgin olive oil
  Interventions: Dietary Supplement: olive oil
- Enriched extra virgin olive oil (Experimental): Enriched extra virgin olive oil
  Interventions: Dietary Supplement: olive oil
- refined olive oil (Placebo Comparator): refined olive oil
  Interventions: Dietary Supplement: olive oil

INTERVENTIONS:
Dietary Supplement: olive oil

SUMMARY:
The present project hypothesizes that the potential protective effect of olive oil relies on its polyphenols profile (quality and quantity) and that it may be synergistic to other food components. Among the nutrients that may be of interest for bone and muscle tissues, unsaturated fatty acids and vitamins are the most described.

Consequently, based on the promising available preliminary data, the present project aims to investigate the possible preventive effect of olive oil polyphenols and eventually the synergistic effects of fatty acids and vitamin D on bone, muscle and adipose tissue, in order to prevent any locomotor dysfunction.

Volunteers will be supplemented during 9 months. The primary and secondary outcome measures will be performed at baseline, 3 and 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian female
* Within at least 7 years post-menopause
* Generally healthy as determined by standard medical assessment on physical and mental health
* Normal weight as determined by BMI (20≤ BMI ≤30)
* Affiliated to National Health Insurance
* Willing to comply with the study procedures
* Willing to accept use of all nameless data, including publication, and the confidential use and storage of all data
* Having received both oral and written explanations about the study
* Having provided her written informed consent

Exclusion Criteria:

* Intestinal or severe metabolic diseases / disorders such as diabetes, renal, hepatic or pancreatic diseases / disorders, ulcer, hyperthyroidism, malignancy, chronic malnutrition
* Osteoporosis (defined by T-score of -2.5 standard deviation (SD) at hip and/or spine)
* On therapy with drugs known to interfere with bone and muscle metabolism
* Taking regular calcium and vitamin D supplements
* Currently participating or having participated in another clinical trial during past 1 year prior to the beginning of this study, this depending on the type of previous study•
* Intense Physical activity

Ages: 57 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2012-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Changes in bone mineral density | at baseline and after 9 months of supplementation

SECONDARY OUTCOMES:
Changes in serum markers of bone resorption | At baseline, 3 and 9 months
changes in serum markers of bone formation | At baseline, 3 and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Coxam, PhD, Study Director — Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Locations (2):
- France (2):
  - Centre de Recherche en Nutrition Humaine, Clermont-Ferrand, Auvergne
  - Centre d'investigation clinique, Marseille, Bouche Du Rhône

REFERENCES:
- See also: Related Info — http://www1.clermont.inra.fr/crnh/